CLINICAL TRIAL: NCT04008498
Title: Amplitude Electroencephalography (aEEG) Monitoring in Preterm Infants: a Feasibility Study on a Neonatal Unit aEEG in Preterm Infants
Brief Title: AEEG in Pre-term Infants
Acronym: AEEG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STH19716
Record Dates: First submitted 2019-04-02; First posted 2019-07-05 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Preterm Infant
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AEEG monitoring (Experimental): Babies whose families consent to involvement will have their head cleaned, EEG leads attached, the monitor set up, and observations.
  Babies will be recorded continuously for the entire duration of their time on the intensive care unit.
  Once the child is receiving high dependency or special care, the investigators will record aEEG for 4 hours once a week until the baby is discharged home. If a participant is moved back to intensive care, the aEEG will be started again if the aEEG monitor is not being used on another baby.
  Before being discharged home, the babies will have additional follow-up. They will receive magnetic resonance imaging (MRI) of the brain on a 1.5T scanner at the University of Sheffield. They will also have a standardised examination of their neurological system performed by a physiotherapist (The Hammersmith Neonatal Neurological Examination).
  Interventions: Diagnostic Test: AEEG brain monitoring

INTERVENTIONS:
Diagnostic Test: AEEG brain monitoring — Babies will be recorded continuously for the entire duration of their time on the intensive care unit.
  Once the child is receiving high dependency or special care, we will record aEEG for 4 hours once a week until the baby is discharged home. If a participant is moved back to intensive care, the aEEG will be started again if the aEEG monitor is not being used on another baby.

SUMMARY:
Amplitude integrated encephalography (aEEG) is a monitor that measures brain activity by attaching leads to a baby's head, and is used routinely in term babies who have brain injury because of a difficult birth. There is little information on how useful aEEG is in premature babies, and most studies only look at small numbers of babies. However, these studies suggest that the aEEG is different in premature babies with brain injury, infections / meningitis, and in those receiving certain drugs. It is also affected by changes in blood pressure and blood acid levels. It is theoretically possible that, if the investigators can detect changes using aEEG early on, the investigators will be able adjust treatment to make a baby better.

DETAILED DESCRIPTION:
At the request of our funder (The Children's Hospital Charity),the investigators have been asked to split the research methodology into two phases to secure the full amount of our funding. The differences between the two phases relates to the length of aEEG recording and whether the babies get the follow-up at discharge from the neonatal unit. The reason for developing two phases is that the funder wishes us to prove the concept that the investigators can recruit premature babies to have aEEG using one machine before they pay for a second monitor to allow for the full study to run. The inclusion and exclusion criteria will be the same for both phases of the study.

PHASE ONE:

Methodology:

The baby of any family who consent to be involved in the study will have their head cleaned using a sterile solution. The 5 sticky EEG leads placed on the head and connected to the monitor. The investigators will not use needle electrodes because of the risk of infection and scarring. The screen of the monitor will be covered with a black piece of card so it is not visible to staff or families. This is because the staff do not know what is a normal or abnormal aEEG in a premature baby, and doctors do not want them making treatment decisions based on a test result they do not understand. However, the investigators will ask the nurses to check the screen at the time of usual observations to check that the monitor is still recording and the leads have not fallen off. This can be done by looking at the "impedance" on the screen, as would happen for babies born at term who have aEEG. Nursing staff will also be asked to review the skin regularly at the time of usual cares to make sure it remains healthy.

The aEEG will be recorded continuously for one week, and will then stop. No further follow-up or intervention is planned.

The funders require us to show proof of concept in 6 premature babies before releasing the remainder of our money for additional monitors, nursing time and equipment.

Staff will review the aEEG monitor at the time of usual observations to ensure that the machine is recording, the impedence is within normal levels, a trace is recorded, the EEG leads remain attached, and the skin condition is good.

PHASE TWO:

Babies whose families consent to involvement will have their head cleaned, EEG leads attached, the monitor set up, and observations as described in phase one. The main difference in the two phases is the timing of recording.

In phase two, babies will be recorded continuously for the entire duration of their time on the intensive care unit.

Once the child is receiving high dependency or special care, the investigators will record aEEG for 4 hours once a week until the baby is discharged home. If a participant is moved back to intensive care, the aEEG will be started again if the aEEG monitor is not being used on another baby.

Before being discharged home, the babies in phase two will have additional follow-up. They will receive magnetic resonance imaging (MRI) of the brain on either a 1.5T or dedicated 3T (Firefly) scanner at the University of Sheffield. They will also have a standardised examination of their neurological system performed by a physiotherapist (The Hammersmith Neonatal Neurological Examination).

The investigators will collect clinical details retrospectively from the observation charts and medical notes, including:

* The gestation age of the baby
* How long they received ventilation or other forms of respiratory support for
* How long they needed oxygen for and, and maximum oxygen requirement each day
* How many infections (sepsis) they had and which organisms were found
* Whether they had a heart defect called a patent ductus arteriosus and whether treatment was needed for this
* What the results of their ultrasound scans of the brain were, which are performed routinely in premature babies
* Whether they had a gut problem called necrotising enterocolitis and whether surgery was needed
* Whether they developed post-haemorrhagic ventricular dilation, and need for intervention
* Survival to discharge

The investigators will ask the families for consent to examine any future medical notes / clinic letters to see what the baby's development was like later in life. The investigators will also ask the families for their permission to contact them in the future in the event that the investigators obtain funding for a follow-on study, such as to examine their child's development in more detail in the future.

The investigators will ask parents to complete a short questionnaire about their experience of the monitoring.

The investigators will ask the neonatal nurses to complete a short questionnaire about their experience of the monitoring and whether they have ideas for improving the process, or any training they would like to have.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants between 26+0 and 30+0 weeks gestational age
* Requiring intensive care following birth
* Live in Sheffield catchment area
* English speaking
* No skin viability issues on the head
* Study aEEG monitor available for use
* No known genetic, congenital structural brain abnormality, congenital infection, metabolic condition or other disorder likely to impact on neurological function independent of preterm birth

Exclusion Criteria:

* Under 26+0 gestational age
* Known genetic, congenital structural brain abnormality, congenital infection, metabolic condition or other disorder likely to impact on neurological function independent of preterm birth
* Non-English speakers
* Non consent

Ages: 26 Weeks to 30 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Recruitment Rate | Upto 24 months after recruitment
  This is a feasibility study to inform the design of a larger multi-centre study. Rate of recruitment will determine how many centre's required for a larger study. Amount of time required to reach recruitment targets will inform average recruitment rate.
Optimal Timing For AEEG Recording | Upto 24 months after recruitment
  This is a feasibility study to inform the design of a larger multi-centre study. The results of full AEEG recordings will demonstrate important time points to be recorded for larger study. Time points of abnormal brain activity will be measured and recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Jessop Wing, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No